CLINICAL TRIAL: NCT05005273
Title: A Phase 2 Randomized Study of BMS-986207 in Combination With Nivolumab and Ipilimumab as First-line Treatment for Participants With Stage IV Non-Small Cell Lung Cancer
Brief Title: A Study to Assess BMS-986207 in Combination With Nivolumab and Ipilimumab as First-line Treatment for Participants With Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA020-016; 2021-000039-29 (EudraCT Number); U1111-1263-4850 (Other: WHO)
Record Dates: First submitted 2021-08-09; First posted 2021-08-13 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; BMS-986207; Nivolumab; Opdivo; Ipilimumab; Yervoy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Drug: BMS-986207
- Arm B (Experimental)
  Interventions: Drug: Nivolumab; Drug: Ipilimumab; Other: Placebo

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-963558
Drug: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
Drug: BMS-986207 — Specified dose on specified days
  Arms: Arm A
Other: Placebo — Specified dose on specified days
  Arms: Arm B

SUMMARY:
The purpose of this study is to determine the safety and efficacy of BMS-986207 in combination with nivolumab and ipilimumab as first-line treatment for participants with stage IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic 1L Stage IV non-small cell lung cancer (NSCLC) of squamous or nonsquamous histology
* No prior systemic anti-cancer treatment given as primary therapy for advanced or metastatic NSCLC
* Measurable disease as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* A formalin-fixed, paraffin-embedded (FFPE) tumor tissue block or a minimum of 20 unstained slides of tumor tissue obtained during screening or prior to enrollment
* Life expectancy of at least 3 months at the time of first dose

Exclusion Criteria:

* Participants with epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or c-ros oncogene 1 (ROS-1) mutations which are sensitive to available targeted inhibitor therapy. Participants with nonsquamous histology and unknown EGFR, ALK, or ROS-1 status are also excluded
* Participants with known B-rapidly accelerated fibrosarcoma proto-oncogene (BRAF) V600E mutations that are sensitive to available targeted inhibitor therapy. Participants with unknown or indeterminate BRAF mutation status are eligible.
* Untreated central nervous system metastases
* Leptomeningeal metastases (carcinomatous meningitis)
* Concurrent malignancy requiring treatment
* Active, known, or suspected autoimmune disease
* Interstitial lung disease
* Uncontrolled or significant cardiovascular disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2022-12-27 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (71):
- United States (17):
  - Local Institution - 0080, Tucson, Arizona
  - Local Institution - 0051, Fountain Valley, California
  - Local Institution - 0070, Fort Myers, Florida
  - Local Institution - 0073, Gainesville, Florida
  - Local Institution - 0036, Orange City, Florida
  - Local Institution - 0045, Pensacola, Florida
  - Local Institution, Port Saint Lucie, Florida
  - Local Institution - 0068, St. Petersburg, Florida
  - Local Institution, Tallahassee, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution - 0081, Boise, Idaho
  - Local Institution - 0077, Coeur d'Alene, Idaho
  - Local Institution - 0074, Edgewood, Kentucky
  - Local Institution - 0002, Ann Arbor, Michigan
  - Local Institution - 0049, Brooklyn, New York
  - Local Institution - 0012, Charleston, South Carolina
  - Local Institution - 0053, Milwaukee, Wisconsin
- Argentina (7):
  - Local Institution - 0009, Pergamino, Buenos Aires
  - Local Institution - 0054, Rosario, Santa Fe Province
  - Local Institution - 0062, Buenos Aires
  - Local Institution - 0021, Buenos Aires
  - Local Institution - 0011, Buenos Aires
  - Local Institution - 0048, Buenos Aires
  - Local Institution - 0057, San Juan
- Australia (3):
  - Local Institution - 0063, Orange, New South Wales
  - Local Institution - 0056, Wahroonga, New South Wales
  - Local Institution - 0052, Warrnambool, Victoria
- Belgium (4):
  - Local Institution - 0034, Mechelen, Antwerpen
  - Local Institution - 0040, Charleroi
  - Local Institution - 0043, Mons
  - Local Institution - 0019, Sint-Niklaas
- Chile (3):
  - Local Institution - 0035, Viña del Mar, Región de Valparaíso
  - Local Institution - 0015, Viña del Mar, Región de Valparaíso
  - Local Institution - 0050, Santiago, Santiago Metropolitan
- France (7):
  - Local Institution - 0037, Limoges
  - Local Institution - 0030, Nantes
  - Local Institution - 0044, Pessac
  - Local Institution - 0016, Rouen
  - Local Institution - 0031, Saint-Priest-en-Jarez
  - Local Institution - 0013, Suresnes
  - Local Institution - 0042, Toulon
- Germany (5):
  - Local Institution - 0005, Gauting, Bavaria
  - Local Institution - 0022, Frankfurt am Main, Hesse
  - Local Institution - 0017, Gera
  - Local Institution - 0023, München
  - Local Institution - 0059, Wiesbaden
- Israel (4):
  - Local Institution - 0064, Haifa
  - Local Institution - 0061, Jerusalem
  - Local Institution - 0078, Jerusalem
  - Local Institution - 0079, Jerusalem
- Italy (5):
  - Local Institution - 0039, Monza, MB
  - Local Institution - 0020, Rozzano, MI
  - Local Institution, Milan
  - Local Institution - 0028, Naples
  - Local Institution - 0001, Padua
- Poland (4):
  - Local Institution - 0024, Bydgoszcz
  - Local Institution - 0003, Lodz
  - Local Institution - 0038, Otwock
  - Local Institution - 0058, Szczecin
- Spain (7):
  - Local Institution - 0033, Majadahonda, Madrid
  - Local Institution - 0041, Alicante
  - Local Institution - 0026, Barcelona
  - Local Institution - 0075, Barcelona
  - Local Institution - 0006, Barcelona
  - Local Institution - 0046, Jaén
  - Local Institution - 0032, Madrid
- Turkey (Türkiye) (5):
  - Local Institution - 0076, Istanbul
  - Local Institution - 0066, Istanbul
  - Local Institution - 0065, Izmir
  - Local Institution - 0067, Samsun
  - Local Institution - 0072, Yüreğir

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant randomized and treated
Groups:
- Treatment 1: nivolumab 360mg Q3W Ipilimumab 1mg/kg Q6W BMS-986207 600mg Q3W
- Treatment 2: nivolumab 360mg Q3W Ipilimumab 1mg/kg Q6W Placebo Q3W
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Study Terminated | 1 | 0

BASELINE CHARACTERISTICS:
Population: 1 participant randomized and treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival by BICR
Description: PFS is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression by BICR or death due to any cause, whichever is earlier.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From first dose to progression or death, 2.3 months
Population: BICR evaluation did not occur so 0 participants were analyzed for this endpoint.
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Progression Free Survival by Investigator
Description: PFS is defined for all randomized participants as the date from randomization to the date of the documentation of disease progression or death due to any cause, whichever is earlier.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From first dose to progression or death, 2.3 months
Population: All Treated Participants
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
Months | 2.3 [NA to NA] — 1 participant analyzed. Lower limit and upper limit cannot be computed via KM methodology. |

3. Secondary Outcome: Overall Response Rate (ORR) by BICR
Description: ORR is defined as the percentage of participants with a confirmed Best overall response of Complete Response (CR) or Partial Response (PR) by RECIST v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to progression or death, 2.3 months
Population: BICR evaluation did not occur so 0 participants were analyzed for this endpoint.
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Overall Response Rate (ORR) by Investigator
Description: as for outcome 3
Time Frame: From first dose to progression or death, 2.3 months
Population: 0 participants met the criteria for to be considered CR and PR, 0 participants were analyzed for this endpoint
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Duration of Response (DOR) by Investigator
Description: DOR is defined for participants who have a confirmed CR or PR as the date from first documented CR or PR per RECIST v1.1 to the date of the documentation of disease progression or death due to any cause, whichever is earlier.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to progression or death, 2.3 months
Population: All Treated Participants
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
Months | NA [NA to NA] — Participant did not meet criteria for CR or PR so could not be evaluated |

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the time of death due to any cause.
Time Frame: From randomization to time of death, 2.3 months
Population: All Treated Participants
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
Months | 2.3 [NA to NA] — only 1 participant treated and analyzed, lower limit number and upper limit number cannot be calculated using KM methodology. |

7. Secondary Outcome: Number of Participants Who Had AEs, SAEs, AEs Leading to Discontinuation and Deaths.
Time Frame: From first dose to progression or death, 2.3 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 1 | 0
Participants
  Adverse Events | 0 | 0
  Serious Adverse Events | 1 | 0
  AEs leading to discontinuation | 0 | 0
  Deaths | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events (From first dose to last dose + 100 days) and All-Cause mortality (From randomization to end of study): 2.3 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Nivolumab 360 mg + Ipilimumab 1 mg/kg + BMS-986207 600 mg: nivolumab 360mg Q3W Ipilimumab 1mg/kg Q6W BMS-986207 600mg Q3W
- Nivolumab 360 mg + Ipilimumab 1 mg/kg + Placebo: nivolumab 360mg Q3W Ipilimumab 1mg/kg Q6W Placebo Q3W
Arm/Group | Nivolumab 360 mg + Ipilimumab 1 mg/kg + BMS-986207 600 mg | Nivolumab 360 mg + Ipilimumab 1 mg/kg + Placebo
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 360 mg + Ipilimumab 1 mg/kg + BMS-986207 600 mg (N=1) | Nivolumab 360 mg + Ipilimumab 1 mg/kg + Placebo (N=0)
Cardiac arrest (Cardiac disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 360 mg + Ipilimumab 1 mg/kg + BMS-986207 600 mg (N=1) | Nivolumab 360 mg + Ipilimumab 1 mg/kg + Placebo (N=0)
Nausea (Gastrointestinal disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to 1 participant being randomized and treated sub group analysis were not completed for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT05005273/Prot_SAP_000.pdf